CLINICAL TRIAL: NCT05893160
Title: Effects of Sustained-release Oral Sodium Nitrite Supplementation on Pain-related Outcomes and Peri- and Postoperative Physiology in People Undergoing Unilateral All-component Revision Total Knee Arthroplasty
Brief Title: Effects of Sustained-release Oral Sodium Nitrite on Postoperative Pain and Recovery Following Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdran per PI's request
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jennifer DeBerry, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300010657; UAB (Other: Anesthesiology)
Record Dates: First submitted 2023-04-12; First posted 2023-06-07 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Intervention (Experimental): The intervention group will receive sodium nitrite SR (40 mg b.i.d. for 30 days)
  Interventions: Drug: JAN101 SR
- Placebo (Placebo Comparator): The comparison group will receive an inert placebo on the same schedule as the intervention group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JAN101 SR — The dosage form of JAN101 to be used in clinical investigations is a sustained release (SR) tablet containing Sodium Nitrite drug substance.
  Other Names: Sodium Nitrite SR
  Arms: Experimental Intervention
Other: Placebo — Inert placebo formulation
  Arms: Placebo

SUMMARY:
This study will determine whether a drug called sodium nitrite helps improve pain and post-operative recovery associated with knee replacement surgery.

DETAILED DESCRIPTION:
The goal of this study is to examine the potential for oral sodium nitrite supplementation to reduce postoperative pain and inflammation and improve functional recovery in individuals undergoing unilateral revision total knee replacement. A sustained release formulation of sodium nitrite (40 mg) administered twice daily will be compared with placebo for a 30-day treatment period. Primary objectives are to evaluate pain and markers of functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals aged 18-70
* Ambulatory with knee pain for greater than 6 months prior to surgery, and willing and able to comply with all study requirements will be considered eligible.

Exclusion Criteria:

* Severe hypertension (systolic blood pressure greater than or equal to 200 mmHg or diastolic blood pressure greater than or equal to 120 mmHg);
* BMI greater than 45 kg/m2;
* Active smoker or stopped smoking within 6 months of enrollment;
* Active local or systemic malignancy, such as lung cancer or leukemia;
* Cardiovascular disease resulting in dyspnea at rest;
* Peripheral neurovascular disease;
* Anemia;
* Hematological disease (eg, coagulopathy, sickle cell disease/anemia);
* Hemoglobin variant;
* Glucose-6-phosphate dehydrogenase deficiency;
* Methemoglobin reductase deficiency;
* Known sensitivity to nitrites;
* Liver disease;
* Use of phosphodiesterase type 5 inhibitors;
* Use of sildenafil (Viagra);
* Systemic treatment with antibiotics, immunosuppressants including corticosteroids, medications for migraine, allopurinol, tricyclic antidepressants, antihistamines, and/or nitrates currently or in the last month;
* Use of nitrovasodilators (e.g. GTN) within the last month;
* Use of protein pump inhibitors within the last month;
* History of substance abuse;
* Recent surgery or hospitalization (within last 6 months);
* Inability to swallow a pill;
* Failure to provide full consent;
* Involvement with a worker's compensation, personal injury, or other legal matter related to participant health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Requirements | 30 days
  Patients
Short-form McGill Pain Questionnaire (SF-MPQ) | 30 days
  The SF-MPQ is a validated test for the measurement of pain. The measure is calculated by summing the point values for responses to 15 questions. Questions 1-11 deal with the sensory dimension of pain (i.e., the quality of the pain). Questions 12-15 deal with the affective dimension of pain (i.e., how the pain affects you). Subscores for the sensory and affective dimensions are calculated, in addition to a total McGill Pain Score. In addition, there is a visual analogue scale for pain and a final question about pain intensity. Higher scores generally correspond to a worse subjective experience of pain.
Brief Pain Inventory (BPI) short form | 30 days
  The BPI is a questionnaire used to assess the severity of pain (intensity) and its impact on functioning (interference). It uses a 0-10 numeric rating scale for item rating and has no scoring algorithm. Pain severity can be measured as the arithmetic mean of the four severity items, with a lower score indicating less pain. Pain interference can be measured from arithmetic mean of the seven interference items, with a lower score indicating less interference.
Pain ratings | 30 days
  Ratings of pain intensity (PI) and pain unpleasantness (PU) will be obtained. A description of the difference between PI (ie, "how strong the pain feels") and PU (ie, "how unpleasant or disturbing the pain is for you") will be read to all participants. Following this, PI and PU will be assessed by asking participants for verbal self-reports on a 0-100 scale, with 0 = "No pain" or "Not at all unpleasant" and 100 = "Pain as intense as I can imagine" or "Pain as unpleasant as I can imagine". Numeric rating scales of PI and PU have demonstrated validity through their ability to detect treatment effects, as well as their strong association with other measures of sensory and affective components of pain.
Quality of Recovery (QoR-15) questionnaire | 30 days
  The QoR-15 scale is a measurement of the quality of recovery from surgery and anesthesia measured in five domains: physical comfort, pain, physical independence, psychological support, and emotional state. The QoR-15 scale provides a score ranging from 0 to 150, with a high score indicating a good quality of recovery.
Physical function | 30 days
  Performance-based measure of physical function will be obtained using a goniometer to measure range of motion (ROM), in degrees from 0-180, at the knee joints. A lower numeric ROM indicates worse physical function.
Leg girth measurement | 30 days
  Girth measurements of both legs will be made while participants are in a reclined position. Knee joint circumference will be measured (in cm), and thigh circumference will be measured (in cm) at 5 cm and 10 cm above the kneecap while thigh muscles are contracted. Measurements will be used to calculate a Limb Symmetry Index ([circumference of injured leg / circumference of uninjured leg] * 100).
White blood cell count | 30 days
  Blood will be drawn for the measurement of white blood cell (WBC) count in # of WBCs per microliter.
Immune cell markers | 30 days
  CD11b/CD18 is a member of the leukocyte integrin family of heterodimeric adhesion molecules expressed on hematopoietic cells and are regarded as immune cell markers. Blood content of CD11b/CD18 expressing cells will be measured using flow cytometry with relative staining and optical density.
Blood markers v1 | 30 days
  Soluble P-selectin, F2-isoprostanes, protein carbonyls, tumor necrosis factor (TNF) alpha, CC chemokine ligand 2 (CCL2), protaglandin E2 (PGE2), and pentraxin 3 (PTX3) will be measured in blood plasma as indices of infection, oxidative stress, and inflammation. They will be quantified in units of pg/ml, where lower levels indicate less infection, oxidative stress, and inflammation.
Blood markers v2 | 30 days
  8-OH-deoxyguanine, nitrate, and nitrite will be measured in blood plasma as indices of oxidative damage and nitric oxide homoeostasis. They will be quantified in micromolar (uM) concentration, where lower levels indicate less oxidative damage.
Timed-Up-and-Go test | 30 days
  This is a test for measuring the functional mobility. Participants will be timed during rising from an armchair, walking 3 meters, turning around, walking back, and sitting down again. Participants will be allowed to use the armrests and will be wearing their shoes.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer DeBerry, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No